CLINICAL TRIAL: NCT07186985
Title: The Effectiveness of Combined Pelvic Floor Muscle Training and Vaginal Oestrogen Therapy in Postmenopausal Women With Stress Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Nguyen Quang Du, Principal Investigator, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMUIRB1843
Record Dates: First submitted 2025-09-09; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Stress Urinary Incontinence (SUI); Postmenopausal Women
Keywords: stress urinary incontinence (SUI); postmenopausal women; Pelvic Floor Muscle Training; Vaginal Oestrogen; Pelvic floor rehabilitation
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor who evaluated participants at baseline, 3 months, and 6 months was blinded and unaware of the participants' intervention group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination of PFMT and vaginal estrogen. (Experimental): Patients were treated with a combination of a pelvic floor rehabilitation program and 0.5 mg vaginal estrogen.
  Interventions: Combination Product: Combined Pelvic Floor Muscle Training and Vaginal Oestrogen Therapy
- vaginal estrogen (Active Comparator): Patients were treated with 0.5 mg topical vaginal estrogen
  Interventions: Drug: Vaginal estrogen

INTERVENTIONS:
Combination Product: Combined Pelvic Floor Muscle Training and Vaginal Oestrogen Therapy — Group 1:
  * Patients were instructed to identify and sense their pelvic floor muscles and to perform contraction-hold-relaxation exercises.
  * Exercises were performed at a frequency of 8 sets per session, 3 sessions per week, progressing from the supine position (month 1), to sitting (month 2), and to standing (month 3). Training was monitored by an electronic diary app. (Appendix)
  * Six individual 45-minute intervention sessions at the center using biofeedback, under the supervision of a physical therapy technician. (Appendix)
  * The training program consisted of two parts: resistance training and pre-contraction training (the Knack technique). (Appendix)
  * Patients were prescribed and instructed to use 0.5 mg vaginal estrogen for 6 months according to the following regimen:
  * First 4 weeks: insert one 0.5 mg tablet nightly at bedtime.
  * Next 20 weeks: insert one 0.5 mg tablet at bedtime twice weekly, with 2-3 days between doses
  Arms: combination of PFMT and vaginal estrogen.
Drug: Vaginal estrogen — Patients were prescribed and instructed to use 0.5 mg vaginal estrogen for 6 months according to the following regimen:
  First 4 weeks: insert one 0.5 mg tablet nightly at bedtime. Next 20 weeks: insert one 0.5 mg tablet at bedtime twice weekly, with 2-3 days between doses.
  Arms: vaginal estrogen

SUMMARY:
The objective of this clinical trial is to investigate whether the combination of pelvic floor muscle training (PFMT) and topical estrogen is more effective in treating stress urinary incontinence (SUI) in postmenopausal women compared to topical estrogen alone. The trial will also analyze factors related to the outcomes of the combined therapy. The key questions this trial aims to answer are:

* Does the combination of PFMT and topical estrogen improve symptoms of stress urinary incontinence in postmenopausal women better than topical estrogen alone?
* Which factors are associated with the effectiveness of the combined therapy?

Researchers will compare the group receiving the combined therapy (pelvic floor muscle training plus topical estrogen) with the group receiving topical estrogen alone to determine whether adding PFMT to estrogen therapy provides additional treatment benefits for SUI in postmenopausal women.

Participants will:

- Be randomly assigned to one of two groups:

Group 1: Undergo a pelvic floor muscle training (PFMT) program combined with topical estrogen therapy (e.g., vaginal cream/application,...).

Group 2: Receive topical estrogen therapy alone (e.g., vaginal cream/application,...).

* Follow the assigned intervention protocol for a specified duration.
* Attend regular clinic visits for clinical examinations, assessment of incontinence severity, and related measurements.
* Monitor and record their incontinence symptoms and the frequency of urine leakage during daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stress urinary incontinence.
* Women who have been naturally postmenopausal for at least 1 year or are postmenopausal due to bilateral oophorectomy (surgical removal of both ovaries).
* Have had sexual intercourse to ensure feasibility of urogenital tract examination and assessment.
* Patients who consent to participate in the study and comply with the treatment protocol, including performing pelvic floor muscle training (PFMT) and completing topical vaginal estrogen therapy.

Exclusion Criteria:

* Patients with concomitant neurological disorders, urinary tract infections, prior pelvic radiotherapy, or congenital malformations of the lower urinary tract.
* Genitourinary malformations or fistulas causing continuous urinary incontinence.
* Genitourinary cancers or tumors of the urinary tract.
* History of spinal cord injury or central nervous system injury affecting the centers that control urination.
* Patients previously treated for stress urinary incontinence (SUI) (surgery, medications, exercises).
* Patients with severe heart disease, coronary artery disease, or myocardial ischemia.
* Patients with pelvic organ prolapse stage III or higher, unexplained vaginal bleeding, confirmed or suspected breast cancer, or vaginitis.
* Presence of premalignant factors or suspected steroid-dependent cancers such as endometrial carcinoma.
* History of or current hepatic tumors, or progressive liver or biliary disease.
* Coagulation/thrombotic disorders, or a history of thromboembolism or stroke.
* Severe hypertriglyceridemia.
* Hypersensitivity to any component of vaginally administered estrogen products.
* The patient or family members are unable to use a smartphone (Android or iOS) to participate in the monitoring program.
* The patient does not agree to participate in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study population consisted of postmenopausal women with stress urinary incontinence
Enrollment: 115 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline at 3 and 6 months in One-hour Pad test | At baseline, 3 months, and 6 months
  One-hour pad test: A noninvasive method that measures the amount of urine leakage collected in an absorbent pad. Standardized by the International Continence Society (ICS), it quantifies leakage during everyday activities, measured in grams (g)

SECONDARY OUTCOMES:
Changes from baseline at 3 and 6 months in Patient Global Impression of Improvement (PGI-I scale) | At baseline, 3 months, and 6 months
  Patient Global Impression of Improvement (PGI-I): Assesses the degree of improvement in urinary incontinence after treatment based on the patient's perception. The scale ranges from "very much better" to "very much worse"
Changes from baseline at 3 and 6 months in International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI-SF scale) | At baseline, 3 months, and 6 months
  International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI-SF scale): Assesses the severity of urinary incontinence and its impact on quality of life, with scores from 0 to 21. Higher scores indicate more severe incontinence
Changes from baseline at 3 and 6 months in Oxford Scale | At baseline, 3 months, and 6 months
  Oxford Scale: Assesses pelvic floor muscle strength, ranging from 0 (no contraction) to 5 (strong contraction)
Changes from baseline at 3 and 6 months in Pelvic floor ultrasound assessment | At baseline, 3 months, and 6 months
  Bladder neck displacement during pelvic floor muscle contraction on ultrasound: Measurement of bladder neck displacement during pelvic floor muscle contraction, in millimeters (mm)
Changes from baseline at 3 and 6 months in Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol scale) | At baseline, 3 months, and 6 months
  Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol scale): Assesses with a total score from 19 to 76 (higher scores reflect worse quality of life)
Changes from baseline at 3 and 6 months in total serum estradiol concentration | At baseline, 3 months, and 6 months
  The concentration of estradiol in serum in all forms, measured in pg/mL